CLINICAL TRIAL: NCT06155825
Title: Nonpharmacological Pain Management in Neonate (A Randomized Controlled Study)
Brief Title: Nonpharmacological Pain Management in Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Mustafaa Abu Zaid, pediatric resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pain management in neonate
Record Dates: First submitted 2023-11-04; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Pain Management; Neonates Pain Management
Keywords: pain management in neonates; nonpharmacological neonatal pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 4 (placebo) (Placebo Comparator): this group will be A control group receive no intervention.
  Interventions: Behavioral: no intervention
- group 1 (interventional group) (Experimental): Intervention groups which will receive nonnutritive suckling.
  Interventions: Drug: nonnutritive suckling
- group 2 (interventional group ) (Experimental): Group 2 will receive oral glucose 25%
  Interventions: Drug: oral glucose 25%
- Group 3 (interventional group) (Experimental): Group 3 will undergo facilitated tuckling
  Interventions: Behavioral: facilitated tuckling

INTERVENTIONS:
Behavioral: no intervention — Group 4 will receive no intervention
  Arms: Group 4 (placebo)
Drug: nonnutritive suckling — Group 1 will receive nonnutritive suckling
  Arms: group 1 (interventional group)
Drug: oral glucose 25% — Group 2 will receive oral glucose 25%
  Arms: group 2 (interventional group )
Behavioral: facilitated tuckling — Group 3 will undergo facilitated tuckling
  Arms: Group 3 (interventional group)

SUMMARY:
This is A randomized controlled study which aim to:

The primary aim in this study is assessment of non-pharmacological pain management in neonate and determine the most effective.

The secondary aim of this study is to introduce idea of neonatal pain management. and record its effect on hospital stay and Duration to reach full enteral feeding. This prospective study will be conducted at NICU unit of Assiut University pediatrician hospital, Duration of study 1 year from 1/12/2023 to 1/12/2024.

one hundred sixty-four children will be divided into 4 groups each group will have 41 patients. Groups 1-3 will be intervention groups, patients of which received a non-pharmacological intervention during mild regular painful maneuvers as cannula insertion, venipuncture, arterial puncture, heel prick, Group 1 will receive nonnutritive suckling. Group 2 will receive oral glucose 25% Group 3 will undergo facilitated tuckling Group 4 will be a control group (receive no nonpharmacological intervention). The pain response in each group will be assessed by CRIES score CRIES comes from (Crying, requires oxygen, Increased vital signs, Expression, Sleep). The scale may be taken over time to monitor the infant's (32 to 60 weeks' gestational age) recovery or response to interventions.

Minimum score is 0 whilst maximum score is 10. The higher the score, the greater the expression of pain. If the CRIES score is greater than 4, further pain assessment should be undertaken, and analgesic administration is indicated for a score of 6 or higher.

DETAILED DESCRIPTION:
Pain is defined as unpleasant sensory and emotional experience associated with tissue damage. Newborns are especially vulnerable to pain and its deleterious effects, as they have larger receptive fields for nociceptive impulses and possibly a higher density of nerve endings and concentration of substance P receptors 1) . The density of proprioceptive nerve ending is equal to the adult, also they have a lower threshold for excitation and sensitization.

In neonates the harmful effects of pain include irritability, fear, sense of mistrust towards caregiver, disturbed sleep and wakefulness cycle, delayed wound healing, altered immunological functions, biochemical alterations in energy metabolism2), negative effects on the developing brain and behavior. Neonates requiring intensive care admission exposed to various types of painful stimuli such as venipuncture, arterial puncture, suction, catheterization or invasive procedures as, lumbar puncture, CVC and bronchoscopy.

The responses to pain in a newborn are nonverbal and include physiological and autonomic manifestations as changes in heart rate, respiratory rate, blood pressure and oxygen saturation3), also behavioral changes as crying, change in facial expressions and body movement. These parameters are used for pain assessment in various scales4). For example, total facial activity and cluster of specific facial findings (brow bulge, eye squeeze, nasolabial furrow, open mouth) were associated with acute and postoperative pain5*6).

Example of most commonly used scales in assessment of pain7), the Premature Infant Pain Profile (PIPP)8), Neonatal Pain Agitation and Sedation Scale (N-PASS)9), Neonatal Infant Pain Scale (NIPS) and the CRIES scale (Crying, Requires Oxygen Saturation, Increased Vital Signs, Expression, Sleeplessness).12)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy term newborn 32 week or more.
2. Newborn during routine painful maneuvers as venipuncture and arterial puncture

Exclusion Criteria:

* 1) Preterm < 32 week 2) Newborn with neurological impairment 3) Sedated newborn 4) Newborn with metabolic diseases 5) Newborn with congenital anomalies 6) Newborn undergoing operative intervention

Min Age: 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
CRIES SCORE | one year
  164 children will be divided into 4 groups each group will have 41 patients. Groups 1-3 will be intervention groups, patients of which received a non-pharmacological intervention during mild regular painful maneuvers as cannula insertion. Group 1,2,3 will be receiving nonpharmacological interventions Group 4 will be a control group. The pain response in each group will be assessed by CRIES score CRIES comes from (Crying, Requires oxygen, Increased vital signs, Expression, Sleep). The scale may be taken over time to monitor the infant's (32 to 60 weeks' gestational age) recovery or response to interventions. Minimum score is 0 whilst maximum score is 10. The higher the score, the greater the expression of pain. If the CRIES score is greater than 4, further pain assessment should be undertaken.

CONTACTS AND LOCATIONS:
Overall Officials: Safaa Mustafaa Abo Zaid, pediatric resident, Principal Investigator — Assiut University; Zeinab Mohie Eldeen, professor, Study Director — Assiut University; Amira Mohamed shalaby, Assistant Professor, Study Director — Assiut University; Randa AbdAlbadea Abdelaleem, Lecturer of Pediatrics, Study Director — Assiut University

REFERENCES:
- [Background] Krechel SW, Bildner J. CRIES: a new neonatal postoperative pain measurement score. Initial testing of validity and reliability. Paediatr Anaesth. 1995;5(1):53-61. doi: 10.1111/j.1460-9592.1995.tb00242.x. PMID 8521311
- [Background] Castagno E, Fabiano G, Carmellino V, Cerchio R, De Vito B, Lauria B, Mercurio G, Coscia A, Ponte G, Bondone C. Neonatal pain assessment scales: review of the literature. Prof Inferm. 2022 Apr 1;75(1):17-28. doi: 10.7429/pi.2022.751017. English, Italian. PMID 36962062
- [Background] Bucsea O, Pillai Riddell R. Non-pharmacological pain management in the neonatal intensive care unit: Managing neonatal pain without drugs. Semin Fetal Neonatal Med. 2019 Aug;24(4):101017. doi: 10.1016/j.siny.2019.05.009. Epub 2019 Jun 5. PMID 31326301
- [Background] Shukla VV, Bansal S, Nimbalkar A, Chapla A, Phatak A, Patel D, Nimbalkar S. Pain Control Interventions in Preterm Neonates: A Randomized Controlled Trial. Indian Pediatr. 2018 Apr 15;55(4):292-296. Epub 2018 Feb 9. PMID 29428919
- [Background] Maxwell LG, Fraga MV, Malavolta CP. Assessment of Pain in the Newborn: An Update. Clin Perinatol. 2019 Dec;46(4):693-707. doi: 10.1016/j.clp.2019.08.005. Epub 2019 Aug 19. PMID 31653303